CLINICAL TRIAL: NCT02508363
Title: Taxi HAILL: A Three-Arm Cluster Randomized Controlled Trial Examining Health Care Access Interventions for Taxi Drivers
Brief Title: Randomized Controlled Trial Examining Health Care Access Interventions for Taxi Drivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: SOUTH ASIAN COUNCIL FOR SOCIAL SERVICES (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-163
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Healthcare Access for Taxi Drivers
Keywords: Taxi drivers; Health care access; 15-163
MeSH Terms: interventions — Surveys and Questionnaires

ARMS (3):
- Health Fair Alone (Control) (Active Comparator): No Follow Up Participant does not require referrals or assistance and was not advised to see a provider in the next three months.
  Regular follow-up call within two weeks of health fair by IHCD intern or staff. Participant has abnormal values, requires referrals or assistance or was advised to see a provider in the next three months.
  Up to 3 call attempts to get participant into needed care. Further contact only by participant request.
  Urgent follow-up call or in-person assistance within 1 day of health fair by IHCD intern or staff Participant advised to seek urgent care within one week.
  Three total call or in-person attempts to get participant into needed care. Further contact only by participant request The follow up call attempts may extend up to 3 months past the date of health fair to complete any needs the driver may have.
  Interventions: Behavioral: questionnaires
- Health Fair + Navigator Case Management (Experimental): • Follow-up call or further in-person assistance within one day for urgent follow-up, or call within two weeks for regular needs. Three call attempts.
  Navigator Case Management by trained staff
  * Tailored assistance for any health needs a minimum of once a month 12 months. Assistance includes pre-appointment reminder calls, post-appointment follow up calls, and health promotion reminders.
  * NCM case management will continue follow-up at a minimum of once per month or as requested by the participant for the study duration and will consistently offer appointment reminders and follow-ups.
  Interventions: Behavioral: questionnaires
- Health Fair + Taxi Health Improvement Promoters (Experimental): Health Fair standard services Follow-up call or further in-person assistance within one day for urgent follow-up, or call within two weeks for regular needs. Three call attempts.
  Taxi health Improvement Promoters (TIPs)
  * Weekly check-ins with each participant, in person or by phone, about scheduling of, and attendance at, primary care appointments along with other health or study questions Mosio Text Messaging Program
  * Send primary care provider recommendations to participant up to three times
  * Two pre-appointment reminders & one post-appointment check-in
  * Twice weekly health promotion reminders after primary care appointment
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires

SUMMARY:
The purpose of this study is to compare the effectiveness of providing the usual health fair service and follow-up alone plus additional interventions of Navigation Case Management (NCM) or mobile text messaging (mTECH) and Taxi health Improvement Promoter (TIP). The addition of NCM or mTECH and TIP to the usual follow-up could prove to be more effective in finding the best way to make sure taxi drivers go to important medical appointments and have a regular doctor to help with their health problems. This study will help researchers find out whether the different approaches are better, the same as, or worse than the usual approach.

In the event that participants are unable to meet in person for biometric measurements, staff will accept their self-reported weight, blood pressure, and waist circumference over the phone. Staff may mail blood pressure machines (to participants who did not receive them at baseline), scales, and measuring tapes to participants to assist in the completion of self-reported biometric measures. Along with supplies, participants may also receive a letter asking for the confirmation of supply receipt.

ELIGIBILITY:
Inclusion Criteria:

Garage/Enrollment Site Inclusion:

* Located in the NYC Borough of Manhattan, Queens, Brooklyn, or the Bronx
* Has a roster of at least 100 drivers or is a site frequented by drivers

Driver Inclusion:

* Male
* Between 21 to 85 years of age (We are selecting participants older than three years past the legal driving age of 18, as younger drivers tend to change jobs more often)
* Planning on remaining in NYC for at least 1 year, (with no vacations or trips to exceed two months)
* Licensed taxi driver for at least three months
* Affillated with a NYC garage or frequents at a study enrollment site
* Speaks English, Bengali, Urdu, Spanish, or French
* Owns a cell phone that can receive text messages and is willing to receive text messages for this study.
* Does not have a usual primary care provider(PCP) at baseline
* Has not seen a doctor for an annual physical within the last year not including annual required physical for work at baseline

TIPs Inclusion:

* Between 21 to 85 years of age
* Male
* Planning on remaining in NYC for at least 1 year, (with no vacations or trips to exceed one month)
* Licensed taxi driver for at least two years
* Affilliated with a NYC garage or frequents at a study enrollment site
* Speaks English, (English proficiency required for TIPs training)
* Willing and able to attend in person TIPs training sessions
* As per study team judgment, based upon the TIPs screening tool, is socially active among fellow taxi drivers, cares about health issues, and wants to help others improve their health

Exclusion Criteria:

Garage/Site Exclusion:

* Does not agree to holding screening health fairs on location (e.g. does not sign enrollment form, or send email confirming agreement, or verbally agree to study team management)

Driver Exclusion:

* Part-time driver (drives fewer than 30 hours per week) Although it is highly unlikely for NYC taxi drivers to work for multiple garages at study baseline, drivers may switch jobs and/or their garage base affiliation while participating in this study. New jobs and/or garage base affiliations will be tracked during follow-up assessments and noted for potential limitations with study retention and intervention contamination. Drivers will be allowed to continue the study even if they are no longer working with the initial garage base.

Ages: 21 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2015-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of drivers that have a primary care provider (pcp) | 12 months
  This primary outcome will be determined through the use of three Medical Expenditure Panel Survey questions (AC05, AC11 and AC22), considered the standard in determining existence of a usual PCP by the AHRQ (11).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Gany F, Narang B, Kakade A, Wu M, Hashemi A, Meraji NN, Li Y, Mehmood R, Acharya S, Leng J. Primary Care Uptake Interventions in Taxi, App-Based, and Other For-Hire Vehicle Drivers: The HAILL Cluster Randomized Controlled Trial. J Gen Intern Med. 2025 May 5. doi: 10.1007/s11606-025-09559-7. Online ahead of print. PMID 40325340
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02508363/ICF_000.pdf